CLINICAL TRIAL: NCT05639413
Title: A Study to Collect Patients, Medical, and Biological Data From Patients Being Treated for Metastatic Colorectal Cancer With a Specific Genetic Mutation: BRAFV600E
Brief Title: A Clinical-biological Prospective Cohort of Patients With BRAFV600E-mutated Metastatic Colorectal Cancer
Acronym: COBRAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UC-GIG-2210/PRODIGE75; 2022-A02232-41 (Other: ID-RCB)
Record Dates: First submitted 2022-11-15; First posted 2022-12-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer; BRAF V600E Mutation Positive
Keywords: Clinical-biological cohort; Colorectal Cancer; BRAF mutation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The COBRAF study was designed as a prospective, multicenter, study. The study is without a therapeutic intervention and is of minimal risk and constraints (category 2 according to the "Loi Jardé"). The study will be conducted in patients with mCRC harboring a BRAFV600E mutation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COBRAF (Other): A 30 mL blood samples (6 mL in each of 5 EDTA tubes) will be collected from each patient at the following timepoints:
  * At the starts of cycle 1, 2 and 3,
  * At 3 and 6 months after starting of each treatment line, if applicable.
  * At disease progression after second-line treatment with encorafenib combined with cetuximab, if applicable.
  * At disease progression after immunotherapy-based treatment in dMMR/MSI patients.
  At most 390 mL of blood will be collected from each patient during the study.
  Interventions: Other: Collection of blood samples

INTERVENTIONS:
Other: Collection of blood samples — A 30 mL blood samples (6 mL in each of 5 EDTA tubes) will be collected from each patient at each timepoint.

SUMMARY:
The study will be conducted in patients with metastatic colorectal cancer (mCRC) harboring a BRAFV600E mutation, to collect clinical data and biological samples to be used for research but also to gather real-world clinical data concerning the treatments and the survival outcomes in patients with this pathology.

DETAILED DESCRIPTION:
Despite substantial progress made in the first- and second line mCRC settings, there are still unmet clinical needs for patients harboring BRAFV600E mutations, especially those with microsatellite stability (MSS) / proficient mismatch repair (pMMR) tumor. The overall survival and access to different treatment in the real-life setting are unknown. Moreover, patient prognosis remains poor and therapeutic resistance to combinations with BRAF inhibitors, is at present, nearly universal. Therefore, it seems essential to prospectively collect clinical and biological data about this rare mCRC subtype. These data will allow us to improve knowledge and to identify clinical and biological factors that could drive therapeutic decisions, predict resistance to treatments, and that are prognostic for survival. In this context, we designed this large, prospective, cohort study to collect clinical data and biological samples to be used for research but also to gather real-world clinical data concerning the treatments and the survival outcomes in patients with BRAFV600E mCRC.

This collection of clinical and biological data (tumor tissue and blood samples) will allow us to identify predictive and prognostic biomarkers with several research work packages planned:

i. To evaluate the circulating tumor DNA (ctDNA) during the metastatic first-, second-, and third-line treatment to:

* Evaluate its positive and negative predictive value.
* Identify molecular alterations preceding and explaining clinical resistance during BRAF/EGFR inhibition therapy and immunotherapy.

ii. To evaluate BRAFV600E mCRC immune environment both at the tumor and blood level (immunomonitoring).

iii. To study specific the dMMR/MSI BRAFV600E subgroup. Furthermore, the data collected will describe the therapeutic management of BRAFV600E mCRC patients in the routine-practice setting which will bring very useful data. The results of the COBRAF study could lay the groundwork to better understand BRAFV600E mCRC and to identify prognostic and predictive biomarkers helping the development of new therapeutic approaches in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years or older
2. Histologically confirmed BRAFV600E metastatic colorectal cancer (mCRC), chemotherapy-naive in the metastatic setting or having initiated a first line of chemotherapy in the metastatic setting (except encorafenib-cetuximab treatment)
3. Available tumor tissue sample obtained before inclusion with sufficient tissue left for biological studies. Patients with only fine-needle aspirations are not eligible.
4. Known MMR/microsatellite status (immunohistochemistry [IHC] and polymerase chain reaction [PCR]) (or under analysis)
5. Patients must have signed a written informed consent form prior to any trial specific procedures. If the patients are physically unable to give their written consent, a trusted person of their choice, not related to the investigator or the sponsor, can confirm in writing the patient's consent.
6. Patients must be willing and able to comply with the study procedures
7. The patient must be affiliated to a social security system or benefit of such a system.

Exclusion Criteria:

1. Patient with another cancer concomitantly with the mCRC requiring treatment or influencing the prognosis according to the medical staff.
2. Patients for whom the follow-up will not be assured by the investigator or its team.
3. Any condition that may jeopardize patient participation in the study as well as non-contraception for men and women with child-bearing potential, and pregnancy or breast feeding for women.
4. Persons deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of first diagnosis of mCRC and the date of death, whatever the cause, up to 5 years
  OS of patients with BRAFV600E mCRC in the real-life setting. The OS is defined as the time between the date of first diagnosis of mCRC and the date of death, whatever the cause. The patients alive at the time of analysis will be censored at the date of their last follow up.

SECONDARY OUTCOMES:
Collection of prospective data about BRAFV600E mCRC | Throughout study completion, up to 5 years
  Prospective collection of data collected during the normal clinical care. A descriptive analysis of the disease (Patients and tumors characteristics), current medical practices (molecular genotyping in France), and therapeutic sequences and composition of each treatment line (patients treated with immunotherapy, patients enrolled in clinical studies, metastatic surgeries). The resulting qualitative data analysis of the population will be expressed in number with percentage.
Correlation between prognostic markers and progression-free survival | From date of first diagnosis of mCRC and date of first progression or death, up to 5 years
  PFS is defined as the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse. PFS will then be correlated to clinical and biological prognostic markers analyzed at date of first diagnosis of mCRC and date of first progression or death by clinical testing used in routine cancer treatment practice (blood test analysis and tumor sample analysis). The Cox proportional-hazards model will then be used to study potential prognostic parameters PFS.
Correlation between prognostic markers and overall survival | Throughout study completion, up to 5 years
  To identify clinical and biological prognostic markers of OS on blood and tumor samples. the OS is defined as the length of time from first diagnosis of mCRC that patients enrolled in the study are still alive. OS will then be correlated to clinical and biological prognostic markers analyzed at date of first diagnosis of mCRC and date of first progression or death by clinical testing used in routine cancer treatment practice (blood test analysis and tumor sample analysis). The Cox proportional-hazards model will then be used to study potential prognostic parameters OS.
Objective response rate | From baseline to first disease progression, up to 5 years
  The objective response rate (ORR) for each treatment line is defined as the percentage of patients with a complete response (CR) or a partial response (PR) for a given treatment line.
Disease control rate | From baseline to first disease progression, up to 5 years
  The disease control rate (DCR) is defined as the percentage of patients with a CR, a PR or stable disease for a given treatment line.
Progression-free survival | From baseline to first disease progression, up to 5 years
  The progression-free survival (PFS) for each treatment line is defined as the time interval between the start of treatment of the given line and the date of the first disease progression (radiological or clinical) or the start of another anticancer therapy, or death from any cause, whichever occurs first.
ctDNA kinetics modeling outcome parameters | From date of first diagnosis of mCRC until the date of first disease progression, up to 5 years
  The detection of ctDNA level assessed by next generation sequencing in the blood of patients with deficient DNA mismatch repair (dMMR) / microsatellite instability (MSI) will be measured at the start of cycle 1, cycle 2, and cycle 3, and at 3 months and 6 months after starting each treatment line, as well as at disease progression.
  The level of ctDNA measured at each time point will provide information on how the body interacts with administered treatments overtime.
Correlation between predictive biomarkers and response to treatment | Throughout study completion, up to 5 years
  These biomarkers of response/resistance to combination treatment with anti-EGFR/anti-BRAF will be assessed by immunohistochemistry analysis of peripheral blood and tumor tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle DE LA FOUCHARDIERE, MD, Principal Investigator — CENTRE LEON BERARD - LYON
Locations (45):
- France (45):
  - Centre Hospitalier D'Avignon, Avignon
  - Centre Hospitalier de Bayeux, Bayeux
  - Chu Simone Veil, Beauvais
  - Institut Bergonie, Bordeaux
  - CH Fleyriat, Bourg-en-Bresse
  - Ch de Cahors, Cahors
  - CH Dr TECHER, Calais
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Chu Estaing de Clermont-Ferrand, Clermont-Ferrand
  - GHPSO, Creil
  - Aphp - Hopital Henri Mondor, Créteil
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Chu de Grenoble Alpes - Hopital Michallon, La Tronche
  - CH Louis Pasteur, Le Coudray
  - Groupe Hospitalier Emile Roux, Le Puy-en-Velay
  - Hopital Franco-Britannique, Levallois-Perret
  - Chu Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Hopital de La Timone, Marseille
  - Intitut Paoli Calmettes, Marseille
  - Grand Hopital de L'Est Francilien - Site de Meaux, Meaux
  - Centre Antoine Lacassagne, Nice
  - CHR d'Orléans, Orléans
  - Aphp - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Aphp - Hopital Bichat, Paris
  - Aphp - La Pitie Salpetriere, Paris
  - Institut Mutualiste Montsouris, Paris
  - Gh Diaconesses Croix Saint Simon, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Ch Perpignan, Perpignan
  - Chu Poitiers, Poitiers
  - Chu de Reims, Reims
  - Chu Rennes Pontchaillou, Rennes
  - Chu de Rouen, Rouen
  - Hôpital Privé de la Loire, Saint-Etienne
  - Hnia Begin, Saint-Mandé
  - Ch de Saint Malo, St-Malo
  - Centre Paul Strauss, Strasbourg
  - Hnia Saint Anne, Toulon
  - Chu de Tours, Tours
  - Chru de Nancy, Vandœuvre-lès-Nancy
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Centre d'Oncologie Saint Yves, Vannes

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.